CLINICAL TRIAL: NCT00339534
Title: Survey of Prostate Cancer in Accra, Ghana
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902240; 02-C-N240
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Prostate Cancer
Keywords: African Men; Case-Control Study; Prostate Cancer; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cases: Cases were recruited at Korle Bu Teaching Hospital in Accra, Ghana, between 2008 and 2012.
- Controls: Controls were selected in a population-based component using a probability sample designed with the 2000 Ghana Population and Housing Census data between 2004 and 2006.

SUMMARY:
This study, conducted at Korle-Bu Hospital in Accra, Ghana, will help elucidate the roles of lifestyle and genetic factors in prostate cancer risk. There is a strong variation in risk of prostate cancer throughout the world. The rates of the disease among African Americans are some of the world s highest. In the United States, the incidence of prostate cancer is 70 percent higher in African Americans than in white Americans and the death rate in African Americans is almost double that of white Americans. The reasons for this excessive risk are unknown, but both genetic and lifestyle factors have been suggested.

Because Africans and African Americans share similar genetic ancestry but have vastly different lifestyles, a better understanding of the rates and risk factor profiles for prostate cancer among Africans will provide important clues to what causes the disease. This study will try to assess the incidence of prostate cancer in the West African nation of Ghana. The study has two components:

* Clinical survey The methods of diagnosis at Korle-Bu will be evaluated and the incidence of prostate cancer over a 5-year period will be estimated.
* Screening and detection survey A survey of 1,000 men between 50 and 74 years of age will estimate the prevalence of both asymptomatic and undiagnosed symptomatic prostate cancer in the Accra population.

The clinical survey will use data from the cancer logbook and medical records at Korle-Bu Hospital and the Ghanaian National Census to derive an estimate of prostate cancer incidence within Accra. The estimate will be low, since it will be based only on men diagnosed or treated at Korle-Bu and will not include men with asymptomatic disease, men diagnosed elsewhere, or men without access to medical care. The screening and detection survey will assess the presence of asymptomatic and unrecognized symptomatic prostate cancer using PSA testing and digital rectal examination in a random sample of 1,000 men in the general population of Accra. This will provide a high estimate of disease prevalence. The two estimates will provide an approximation of the true incidence rate of the disease in Accra.

Comparison of these data with similar data from community surveys of African Americans will provide insight into reasons for the excess risk of prostate cancer in African Americans.

DETAILED DESCRIPTION:
OBJECTIVE: The key aim of this study is to assess the burden of prostate cancer in Ghana and to evaluate how the impact of prostate cancer among West Africans compares with that among African Americans, whose reported incidence rates are among the highest in the world. West Africans and African Americans share genetic ancestry but have very different lifestyles and environmental exposures. The study aim will be achieved by establishing lower and upper bounds on the true incidence of prostate cancer in the capital city of Accra. The secondary aim of the study is to establish epidemiological, biochemical, and genetic profiles of West Africans for comparisons with African Americans to provide etiologic clues for prostate cancer. DESIGN: The study will consist of two components: 1. a clinical survey, a. divided into a five-year retrospective, and b. a 3-year prospective phase, and 2. a population screening survey.

ELIGIBILITY:
* INCLUSION CRITERIA:

The 1,000 Accra residents selected for screening will include 300 men 50-59, 400 men 60-69, and 300 men 70-74 years of age.

EXCLUSION CRITERIA:

Men who do not meet the age requirements will be excluded from the study.

In addition, men who have a history of prostate cancer for which they have received treatment will also be excluded (men with untreated prostate cancer will be included).

Ages: 18 Years to 125 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for analysis were recruited through the Ghana Prostate Study-a population-based component, and a clinical component. The population-based component was a probability sample designed using the 2000 Ghana Population and Housing Census data which successfully recruited 1,037 healthy men between 2004 and 2006. Consented individuals underwent an in-person interview, and within 7 days had a digital rectal examination (DRE) and provided an overnight fasting blood sample for PSA testing, biomarker assays, and genetic analysis. Subjects who had a positive screen by PSA ([2.5 ng/ml) or DRE underwent a transrectal ultrasound-guided biopsy. A total of 73 histologically confirmed prostate cancer cases were identified through the population-based screening component of the Ghana Prostate Study. We also recruited 676 prostate cancer cases at Korle Bu Teaching Hospital in Accra, Ghana, between 2008 and 2012.
Sampling Method: Probability Sample
Enrollment: 1758 (Actual)
Dates: Start 2002-06-26 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Prostate cancer | At recruitment: case-control study
  Prostate cancer (case-control observational/epidemiologic study)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Cook, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Ghana Medical-Korle Bu Teaching Hospital, Accra, Ghana